CLINICAL TRIAL: NCT02049021
Title: Pilot Double Blind, Placebo Controlled and Randomized Study to Assess Electroconvulsive Therapy Efficacy as Augmenting Strategy to Clozapine in Super-refractory Schizophrenia
Brief Title: Electroconvulsive Therapy (ECT) in Patients With Super Refractory Schizophrenia
Acronym: SSURECT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Helio Elkis, MD, PhD ; Associated Professor of the Departament of Psychiatric, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ECT Schizo
Record Dates: First submitted 2014-01-15; First posted 2014-01-29 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Refractory Schizophrenia; Super Refractory Schizophrenia
Keywords: schizophrenia; electroconvulsive therapy; refractory Schizophrenia; super refractory schizophrenia; clozapine
MeSH Terms: conditions — Schizophrenia, Treatment-Resistant; Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electroconvulsive Therapy (Experimental): Patients in use of clozapine randomized to receive ECT treatment
  Interventions: Device: MECTA SPECTRUM 5000Q ECT
- SHAM ECT (Sham Comparator): Patients receiving clozapine randomized to sham ECT (placebo)
  Interventions: Procedure: Sham ECT

INTERVENTIONS:
Device: MECTA SPECTRUM 5000Q ECT
  Other Names: ECT; Electrochock; electroconvulsive therapy device
  Arms: Electroconvulsive Therapy
Procedure: Sham ECT — Sedation using propofol or etomidate and usual ECT preparation (no stimulation)
  Arms: SHAM ECT

SUMMARY:
Introduction: In spite of recent advances in schizophrenia treatment, 30% of patients still do not respond properly to antipsychotic therapy. These patients are considered treatment-resistant or refractory, and the best choice for them is clozapine. However, even supported by the literature as the best known antipsychotic in terms of efficacy and rates of response, a considerable number of patients will still not respond to this treatment, remaining symptomatic and dysfunctional. These patients are classified as super-refractory (clozapine-resistent). In these cases, augmenting strategies are necessary, and some have been in use: typical and atypical antipsychotics, mood stabilizers, antidepressants and electroconvulsive therapy (ECT). Some studies have favored ECT, but no definitive conclusion has been drawn.

Objective: Test the electroconvulsive therapy efficacy and safety as augmenting strategy to clozapine-resistant patients, as compared to placebo (sham ECT).

Methods: This is a pilot double blind, placebo controlled and randomized study to assess electroconvulsive therapy efficacy as augmenting strategy to clozapine in super-refractory schizophrenia. The ECT treatment will be delivered with either a MECTA SPECTRUM 5000Q or 4000Q device, and the procedure is under general anesthesia and monitorization, after informed consent. The Hospital will follow national protocols and regulations on ECT. Sham ECT consists in habitual patient preparation and sedation, without stimulation. Patients that fit inclusion criteria will have their clozapine blood levels dosed and undergo structured assessments at baseline, after 6 treatments and at the end of the cycle of 12 ECT sessions (thrice a week protocol). The assessments will be based on CGI (Clinical Global Impression) and PANSS (Positive and Negative Syndrome Scale) scales. All medication will be maintained, except lithium carbonate.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia or schizoaffective disorder (DSM-IV-TR);
* Ages between 18 and 55 years old, both genders;
* Must be using adequate contraception if a fertile woman;
* Must be on clozapine treatment for at least 6 months, with or without augmenting strategies;
* Must be clozapine-resistent (super-refractory patient), defined by a CGI-severity ≥ 4, PANSS total score ≥ 60 and at least 4 items of the positive subscale ≥ 4 at baseline.

Exclusion Criteria:

* Clinical somatic disease not stabilized in the three months preceding the study;
* Other Axis I disorders (DSM-IV-TR);
* Laboratory tests with significantly abnormal values that persist for more than two weeks;
* Lack of permanent residence during the study period;
* History of poor treatment adherence.
* History of ECT use in the past six months that precede the start of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-02; Primary Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
PANSS change from baseline | 4 weeks
  Structured assessments will be done at baseline, and at the end of the cycle of 12 ECT sessions (thrice a week protocol). The assessments will be based on PANSS (Positive and Negative Syndrome Scale). Changes from Baseline on this scale will be documented after a 4 weeks period.
PANSS change from baseline | 2 weeks
  Structured assessments will be done at baseline, and at the end of the cycle of 6 ECT sessions (thrice a week protocol). The assessments will be based on PANSS (Positive and Negative Syndrome Scale). Changes from Baseline on this scale will be documented after a 2 week period.

SECONDARY OUTCOMES:
CGI change from baseline | 4 weeks
  Clinical Global Impression will be assessed as well, along with PANSS scale, and changes compared to baseline.
CGI change from baseline | 2 weeks
  Clinical Global Impression will be assessed as well, along with PANSS scale, and changes compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Hélio Elkis, MD PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Institute of Psychiatry - Clinics Hospital - University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Elkis H. Treatment-resistant schizophrenia. Psychiatr Clin North Am. 2007 Sep;30(3):511-33. doi: 10.1016/j.psc.2007.04.001. PMID 17720034
- [Background] Havaki-Kontaxaki BJ, Ferentinos PP, Kontaxakis VP, Paplos KG, Soldatos CR. Concurrent administration of clozapine and electroconvulsive therapy in clozapine-resistant schizophrenia. Clin Neuropharmacol. 2006 Jan-Feb;29(1):52-6. doi: 10.1097/00002826-200601000-00012. PMID 16518135
- [Background] Kho KH, Blansjaar BA, de Vries S, Babuskova D, Zwinderman AH, Linszen DH. Electroconvulsive therapy for the treatment of clozapine nonresponders suffering from schizophrenia--an open label study. Eur Arch Psychiatry Clin Neurosci. 2004 Dec;254(6):372-9. doi: 10.1007/s00406-004-0517-y. Epub 2004 Nov 12. PMID 15538604
- [Background] Lehman AF, Lieberman JA, Dixon LB, McGlashan TH, Miller AL, Perkins DO, Kreyenbuhl J; American Psychiatric Association; Steering Committee on Practice Guidelines. Practice guideline for the treatment of patients with schizophrenia, second edition. Am J Psychiatry. 2004 Feb;161(2 Suppl):1-56. No abstract available. PMID 15000267
- [Background] Miller A, Hall CS, Buchanan RW, Buckley PF, Chiles JA, Conley RR, Crismon ML, Ereshefsky L, Essock SM, Finnerty M, Marder SR, Miller DD, McEvoy JP, Rush AJ, Saeed SA, Schooler NR, Shon SP, Stroup S, Tarin-Godoy B. The Texas Medication Algorithm Project antipsychotic algorithm for schizophrenia: 2003 update. J Clin Psychiatry. 2004 Apr;65(4):500-8. doi: 10.4088/jcp.v65n0408. PMID 15119912
- [Background] Tang WK, Ungvari GS. Efficacy of electroconvulsive therapy in treatment-resistant schizophrenia: a prospective open trial. Prog Neuropsychopharmacol Biol Psychiatry. 2003 May;27(3):373-9. doi: 10.1016/S0278-5846(02)00354-8. PMID 12691772
- [Background] Tharyan P, Adams CE. Electroconvulsive therapy for schizophrenia. Cochrane Database Syst Rev. 2002;(2):CD000076. doi: 10.1002/14651858.CD000076. PMID 12076380
- See also: Institute of Psychiatry - University of Sao Paulo — http://www.ipqhc.org.br/
- See also: Department of Psychiatry - University of Sao Paulo Medical School — http://www.psiquiatriafmusp.org.br/departamento/